CLINICAL TRIAL: NCT01429896
Title: The Effect of Extrinsic Factors on Food Allergy
Acronym: Ex-Factor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: Imperial College London (Other); University of Manchester (Other)
Responsible Party: Principal Investigator, Dr. Andrew Clark, Associate Lecturer and Consultant in Paediatric Allergy, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 01.31.09.2011
Record Dates: First submitted 2011-08-31; First posted 2011-09-07 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Peanut Hypersensitivity
Keywords: peanut allergy; food allergy; thresholds; anaphylaxis; food labelling; food challenges; peanut challenges
MeSH Terms: conditions — Peanut Hypersensitivity; Food Hypersensitivity; Anaphylaxis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Arm 1 (Experimental): Exercise followed by sleep restriction followed by control challenge
  Interventions: Other: Food challenge
- Arm 2 (Experimental): Sleep restriction followed by exercise followed by control challenge
  Interventions: Other: Food challenge
- Arm 3 (Experimental): control followed by sleep restriction followed by exercise
  Interventions: Other: Food challenge
- Arm 4 (Experimental): control followed by exercise followed by sleep restriction
  Interventions: Other: Food challenge
- Arm 5 (Experimental): Sleep Restriction followed by control followed by exercise
  Interventions: Other: Food challenge
- Arm 6 (Experimental): Exercise followed by control followed by sleep restriction
  Interventions: Other: Food challenge

INTERVENTIONS:
Other: Food challenge — Double blind placebo controlled peanut challenge. Each challenge given with or without extrinsic factors exercise or sleep restriction.
  Other Names: Threshold extrinsic factor challenges

SUMMARY:
Food allergy is a common problem, affecting 5-8% of the population. Peanut allergy causes reduced quality of life due to the perceived high risk of severe reactions. Patients rely on accurate labeling of both loose and pre-packed foods, but these are often ambiguous and unhelpful. There is a common conception that labeling is 'over-cautious'. Peanut-allergic consumers face increasingly restricted food choices in complying with this advice due, in part, to the proliferation of advisory labels such as 'may contain peanuts'. This contributes to the reduces quality of life of affected individuals.

For industry to provide more accurate and helpful labeling, certain characteristics of the food-allergic population need to be defined. Firstly, the minimum 'eliciting dose' for the population has been estimated by studying large groups of peanut allergic patients who are challenged with peanut ingestion in increasing amounts. From these, an eliciting dose that provokes a reaction in 10% of the food-allergic population has been estimated at between six and 14mg of peanut protein.

Translation of population eliciting doses (ED) into acceptable levels of allergen contamination for the population requires consideration of a 'safety factor'- to account for individual variability in dose threshold and severity. Data suggest such variability depends in part on extrinsic factors (exercise and sleep restriction). Each factor may have a different effect in scale and direction. The investigators are proposing a cross-over trial with 85 peanut-allergic adults who will each undergoing a baseline peanut challenge followed by repeat challenges with extrinsic factors applied, in random order (repeat baseline, +exercise and +sleep restriction). These data will further define ED for the UK population and a safety factor derived from shift in threshold, to inform industry and protect the allergic population.

DETAILED DESCRIPTION:
N=100 subjects will undergo a baseline challenge to peanut without exacerbating extrinsic factors. These initial baseline challenges will be performed when asthma is well controlled (validated by normal spirometry values), the subject is rested and there is no evidence of viral illness (clinical history and examination). A two-day double blind placebo controlled peanut challenge (DBPCPC) will be performed. Subjects receive either all placebo doses or all active doses on one of two days. Each day consists of all eight doses separated by 20 minute intervals (3microg to 1g). The active doses are hidden in a carrier which has been assessed for blinding efficacy. Subjective and objective dose threshold and severity score for challenge outcome will be recorded. Subjects will receive detailed written and verbal advice to avoid peanut until the next challenge. All subjects will be asked to carry oral antihistamines and injectable adrenaline.

All participants who have a clinical reaction during the initial baseline DBPCFC will be randomized to one of 6 balanced cross over intervention sequences from a Latin square design. Each group rotates through three further challenges in a different order: control (no extrinsic factor), exercise and sleep restriction.

1. Control challenge

   Subjects must not have had any accidental reaction to peanut in the previous three months. This challenge will be performed when asthma is well controlled (validated by spirometry normal values), the subjects are rested (sleep diary for preceding week will be examined) and there is no viral illness (clinical history and examination). A peanut challenge will be performed (identically to the initial baseline DBPCFC). Dose threshold and severity score for challenge outcome will be recorded.
2. Exercise challenge Subjects undergo a repeat challenge to peanut with exercise as an extrinsic factor, a minimum of three months after the previous challenge. Subjects must not have had any accidental reaction to peanut in the previous three months. This challenge will be performed when asthma is well controlled (validated by spirometry normal values for the individual and clinical history), the subjects are rested, and there is no viral illness.

The challenge will be double blind and placebo controlled. The challenge will take place on two occasions, on one day all four doses will contain placebo only, on the second all four doses will be active (peanut). The subjects will undergo an identical exercise protocol on both days.

On each day the challenge will begin with 15 minutes of exercise using a standardised protocol. Following this the first challenge dose is given. This is followed by 20 minutes of rest (and observation) before a further exercise period followed by ingestion of the second dose and so on.

The active doses will be…

1. 1/100th of the threshold identified at the initial baseline challenge
2. 1/10th of the threshold identified at the initial baseline challenge
3. The threshold dose identified at the control challenge
4. One dose increment higher than the dose identified at the control challenge.

Subjective and objective dose thresholds and severity score for challenge outcome will be recorded.

If there is no reaction to any dose on the active day then the active arm will be repeated on a separate day, starting at the lowest available challenge dose (3 micrograms). Dose increments up to at least 1/100th of the threshold identified at the control challenge will follow.

3. Sleep restriction

Participants will undergo a repeat double blind placebo controlled challenge to peanut including sleep restriction as an extrinsic factor, a minimum of three months from the last challenge. Subjects must not have had any accidental reaction to peanut in the previous three months. This challenge will be performed when asthma is well controlled (validated by spirometry normal values), and there is no viral illness (clinical history and examination).

Subjects will be admitted to the research ward on the evening prior to the challenge. Overnight, sleep will be restricted to 3 hours (2300-0200). Subjects will undergo a peanut challenge, using the same dosing range and intervals as the initial baseline challenge.

Subjective and objective dose thresholds and severity score for challenge outcome will be recorded on central online data store. The challenge will take place on two occasions, on one day all doses will contain placebo only, on the second all doses will be active (peanut). The subjects will undergo an identical sleep restriction protocol on each day.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed.
* Male and female subject who are 18-45 years of age at the time of study entry (Visit 1) who have a diagnosis of acute peanut allergy as manifested by urticaria, angioedema or respiratory/gastrointestinal tract symptoms, with acute onset of symptoms after ingestion (up to 2h).
* A positive peanut DBPCFC at baseline (Visit 1). This outcome is defined as the onset of objective allergic events after ingestion of peanut protein but not to the placebo. Eligibility to the DBPCFC requires fulfillment of all other eligibility criteria at visit 1.
* Subjects must be able to comply with the study procedures.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-09 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
minimum amount of peanut protein in milligrams which causes an objective clinical reaction during peanut challenges | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T Clark, MB BS MD, Study Director — Cambridge University Hospitals NHS Trust
Locations (2):
- United Kingdom (2):
  - Addenbrooke's Hospital, Cambridge, Cambs
  - Imperial College, London, London

REFERENCES:
- [Background] Avery NJ, King RM, Knight S, Hourihane JO. Assessment of quality of life in children with peanut allergy. Pediatr Allergy Immunol. 2003 Oct;14(5):378-82. doi: 10.1034/j.1399-3038.2003.00072.x. PMID 14641608
- [Derived] Dua S, Ruiz-Garcia M, Bond S, Durham SR, Kimber I, Mills C, Roberts G, Skypala I, Wason J, Ewan P, Boyle R, Clark A. Effect of sleep deprivation and exercise on reaction threshold in adults with peanut allergy: A randomized controlled study. J Allergy Clin Immunol. 2019 Dec;144(6):1584-1594.e2. doi: 10.1016/j.jaci.2019.06.038. Epub 2019 Jul 15. PMID 31319102